CLINICAL TRIAL: NCT00562367
Title: Biochemical Brain Changes Correlated With The Antidepressant Effect Of Thyroid Hormones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2001-P-000836
Record Dates: First submitted 2007-11-20; First posted 2007-11-22 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Triiodothyronine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cytomel (liothyronine) — Cytomel (liothyronine) 25-50 mcg/day for 4 weeks

SUMMARY:
We propose to investigate structural and biochemical brain abnormalities in depressed subjects, and the relationship between the presence of such abnormalities and treatment outcome. We will recruit N=20 subjects with major depression disorder and N=20 matched normal controls. The depressed subjects would have previously not responded to an adequate trial with a selective serotonin reuptake inhibitor (SSRI). These depressed subjects will be treated for 4 weeks with the same SSRI antidepressant and with adjuvant triiodothyronine (T3). Structural magnetic resonance images (MRI) and then Phosphorus-31 magnetic resonance spectroscopic imaging (31P-MRSI) data will be obtained two times for each patient (at the beginning and at the end of the study) and one time for the normal controls. We will measure for each depressed subject the number of white matter hyperintensities (WMH); we will also measure the degree of change from baseline in several compounds characteristic for the cellular high-energy phosphate metabolism: the phosphocreatine/inorganic phosphate ratio and the beta-nucleoside triphosphate. We will compare the severity of WMH and the high-energy phosphate metabolism in two groups of depressed subjects (those responding and those not responding to thyroid hormone augmentation) and the normal controls.

We hypothesize that:

1. All depressed subjects, when compared with normal controls, will present lower baseline levels of compounds characteristic for the high-energy phosphate metabolism.
2. Depressed subjects responding to T3 augmentation, when compared with subjects not responding to T3 augmentation, will present a larger increase of the high-energy phosphate metabolism.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnostic criteria for MDD (diagnosed with the use of SCID)
* Written informed consent
* Men or women aged 18-65
* A baseline Hamilton-D17 score of > 16.

Exclusion Criteria:

* Subjects with suicidal ideation where outpatient treatment is determined unsafe by the study clinician. These patients will be immediately referred to appropriate clinical treatment.
* Pregnant women or women of childbearing potential who are not using a medically accepted means of contraception (defined as oral contraceptive pill or implant, condom, diaphragm, spermicide, IUD, s/p tubal ligation, partner with vasectomy)
* Serious or unstable medical illness, including cardiovascular, hepatic, renal, respiratory, endocrine, neurologic or hematologic disease
* History of seizure disorder,
* History or current diagnosis of the following DSM-IV psychiatric illness: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, patients with mood congruent or mood incongruent psychotic features, patients with substance dependence disorders, including alcohol, active within the last 12 months.
* History or current diagnosis of dementia, or a score of < 26 on the Mini Mental Status Examination (Folstein, 1975) at the screening visit.
* History of multiple adverse drug reactions or allergy to the study drugs.
* Patients with mood congruent or mood incongruent psychotic features.
* Patients having shown minimal or no response to a standard course of antidepressant treatment with an SSRI. A standard course will be defined as the following medications taken for > 4 weeks: fluoxetine > 20 mg/day, sertraline > 50 mg/day, paroxetine > 20 mg/day, fluvoxamine > 50 mg/day, citalopram > 20 mg/day, venlafaxine > 150 mg/day.
* Clinical or laboratory evidence of hypothyroidism.
* Patients who have had electroconvulsive therapy (ECT) within the 6 months preceding baseline.
* History of intolerance to Cytomel
* History of cardiac pathology or diabetes

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2001-10; Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
change in depression (as measured by Ham-D-17) over the 4 weeks study | 4 weeks

SECONDARY OUTCOMES:
change in bioenergetic metabolism (e.g., NTP and PCr) as measured by phosphorus magnetic resonance spectroscopy (P31-MRS) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dan V Iosifescu, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Iosifescu DV, Nierenberg AA, Mischoulon D, Perlis RH, Papakostas GI, Ryan JL, Alpert JE, Fava M. An open study of triiodothyronine augmentation of selective serotonin reuptake inhibitors in treatment-resistant major depressive disorder. J Clin Psychiatry. 2005 Aug;66(8):1038-42. doi: 10.4088/jcp.v66n0812. PMID 16086620
- [Derived] Iosifescu DV, Bolo NR, Nierenberg AA, Jensen JE, Fava M, Renshaw PF. Brain bioenergetics and response to triiodothyronine augmentation in major depressive disorder. Biol Psychiatry. 2008 Jun 15;63(12):1127-34. doi: 10.1016/j.biopsych.2007.11.020. Epub 2008 Jan 22. PMID 18206856